CLINICAL TRIAL: NCT01406002
Title: An Open-label, One-sequence Study to Evaluate the Effect of Multiple Doses of Rifampicin on the Pharmacokinetics of YM150 (Darexaban) and Metabolites in Young Healthy Male Subjects
Brief Title: To Evaluate if Multiple Doses of Rifampicin Change the Blood Concentration of YM150 (Darexaban)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 150-CL-045; 2009-015763-13 (EudraCT Number)
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-03

CONDITIONS: Pharmacokinetics of Darexaban and Metabolites; Healthy Subjects
Keywords: Pharmacokinetics; darexaban; YM150; rifampicin; Phase 1
MeSH Terms: interventions — darexaban; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm 1 (Experimental): darexaban, wash-out, rifampicin + darexaban
  Interventions: Drug: darexaban; Drug: Rifampicin

INTERVENTIONS:
Drug: darexaban — oral
  Other Names: YM150
Drug: Rifampicin — oral
  Other Names: Rifadin

SUMMARY:
The primary objective of this study is to determine the effect of rifampicin on the way the body handles darexaban and its metabolites (drug degradation products). The secondary objective of the study is to evaluate the safety and tolerability of a single dose of darexaban alone and when administered together with rifampicin.

DETAILED DESCRIPTION:
This is an open-label, 1-sequence study in young healthy male subjects to evaluate the effect of multiple daily doses of rifampicin on the PK of darexaban and metabolites after a single dose of darexaban. In addition, safety and tolerability of darexaban administered alone and in combination with rifampicin is evaluated. Eligible subjects are admitted to the clinical unit in the morning of Day -1.

Subjects receive a single dose of darexaban on Day 1. Subjects then receive rifampicin once daily (qd) on Days 4-14.On Day 11, the second single dose of darexaban is given in combination with rifampicin.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.5-30.0 kg/m2
* Male subjects must be non-fertile, i.e. surgically sterilized or must practice an adequate contraceptive method to prevent pregnancies

Exclusion Criteria:

* Known or suspected hypersensitivity to darexaban or rifampicin or any components of the formulation used
* Any of the liver function tests (i.e. ALT and AST) above the upper limit of normal at repeated measures
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic as judged by the medical investigator
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests
* Use of any prescribed or OTC drugs (including vitamins, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior to admission to the Clinical Unit, except for occasional use of paracetamol (up to 3 g/day)
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampicin) in the 3 months prior to admission to the Clinical Unit
* Any use of drugs of abuse, or smoking of more than 10 cigarettes (or equivalent) or more than 21 units (210 g) of alcohol per week within the 3 months prior to study Donation of blood or blood products within 3 months prior to admission to the Clinical Unit
* Participation in any clinical study within 3 months or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study, provided that the clinical study did not entail a biological compound with a long terminal half life

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of darexaban and its metabolites assessed by plasma concentration | Plasma samples are taken until 72 hours after darexaban dosing

SECONDARY OUTCOMES:
Monitoring of safety and tolerability through assessment of vital signs, ECG, clinical safety laboratory and adverse events | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.; Prinicpal Investigator, Principal Investigator — SGS Aster, Paris, France
Locations (1):
- SGS Aster, Paris, France

REFERENCES:
- [Background] Groenendaal D, Strabach G, Garcia-Hernandez A, Kadokura T, Heeringa M, Mol R, Eltink C, Onkels H. The pharmacokinetics of darexaban are not affected to a clinically relevant degree by rifampicin, a strong inducer of P-glycoprotein and CYP3A4. Br J Clin Pharmacol. 2013 Feb;75(2):440-9. doi: 10.1111/j.1365-2125.2012.04346.x. PMID 22642721